CLINICAL TRIAL: NCT02722525
Title: Impact of Anti-androgen Treatment on Cardiac Function
Brief Title: Cardiac MRI in Measuring the Impact of Anti-androgen Treatment on Cardiac Function in Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Pelontonia (Unknown)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-14186; NCI-2015-00029 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-11-18; First posted 2016-03-30 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Injury; Prostate Carcinoma
Keywords: ADT; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (cardiac MRI, skeletal muscle PMRS) (Experimental): Patients undergo a treadmill stress CMR focused on cardiac muscle comprised of resting MRI over 10-15 minutes followed by treadmill exercise until peak stress. Patients then undergo MRI and gadopentetate dimeglumine perfusion imaging immediately after exercise and after a 6-8 minute recovery period. Within 24 hours of treadmill CMR exam, patients also undergo skeletal muscle PMRS while at rest, during, and in the recovery phase of resistive lower extremity exercise which patients complete over 30 seconds. Both procedures are performed before initiation of ADT treatment (baseline) and 4-7 months after initiation of ADT treatment.
  Interventions: Procedure: Magnetic Resonance Imaging; Behavioral: Exercise Intervention; Procedure: Perfusion Magnetic Resonance Imaging; Procedure: Spectroscopy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo treadmill stress CMR
  Other Names: Magnetic Resonance Imaging Scan; MRI; MRI Scan; NMRI
Behavioral: Exercise Intervention — Complete treadmill exercise
Procedure: Perfusion Magnetic Resonance Imaging — Undergo gadopentetate dimeglumine perfusion MRI
  Other Names: PW-MRI
Behavioral: Exercise Intervention — Complete resistive lower extremity exercise
Procedure: Spectroscopy — Undergo skeletal muscle PMRS
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Learning about the impact of anti-androgen treatment has on cardiac function in patients with prostate cancer may help plan treatment and help patients live more comfortably. This pilot clinical trial will utilize cardiac magnetic resonance imaging (MRI) before a patient starts hormone therapy and after 4 to 7 months of hormone therapy. The objective is to measure the impact of hormone therapy (anti-androgen treatment) on cardiac function in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the impact of a minimum of 4 months of full androgen deprivation therapy (ADT) on cardiac and skeletal muscle structure and performance using novel cardiovascular magnetic resonance (CMR) approach.

OUTLINE:

Study participants will undergo a treadmill stress CMR focused on cardiac muscle comprised of resting MRI over 10-15 minutes followed by treadmill exercise until peak stress. Patients then undergo MRI and gadopentetate dimeglumine (Gd-diethylenetriamine penta-acetic acid [DTPA]) perfusion imaging immediately after exercise and after a 6-8 minute recovery period. Within 24 hours of treadmill CMR exam, patients also undergo skeletal muscle phosphorus magnetic resonance spectroscopy (PMRS) while at rest, during, and in the recovery phase of resistive lower extremity exercise which patients complete over 30 seconds. Both procedures are performed before initiation of ADT treatment (baseline) and 4-7 months after initiation of ADT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have biopsy proven carcinoma of the prostate
* Be planning to begin a course of at least 4 months of ADT; the ADT is defined as: (a) surgical castration; (b) gonadotropin-releasing hormone (GNRH) antagonist alone; (c) GNRH antagonist with oral androgen receptor blockade, and (d) GNRH antagonist, oral androgen receptor blockade, and 5-alpha reductase inhibitors; we will not include men with only oral anti-androgen therapy such as 5-alpha reductase inhibitors alone or oral anti-androgens alone
* Have an ECOG (Eastern Cooperative Oncology Group) performance status of 0-1
* Have plasma total cholesterol < 200 mg/dL
* Have plasma triglycerides < 200 mg/dL
* Have BUN/Cr (Blood urea nitrogen and serum creatinine) without clinically significant abnormalities after review by the study physicians
* Liver enzymes without clinically significant abnormalities after review by the study physicians
* CBC (complete blood count) without clinically significant abnormalities after review by the study physicians
* PT/PTT/INR (prothrombin time/partial thromboplastin time) without clinically significant abnormalities after review by the study physicians
* Voluntarily agree to participate and sign an informed consent document

Exclusion Criteria:

* Have an active malignancy other than prostate cancer that requires therapy
* Not be undergoing evaluation and workup for active cardiovascular disease; men with treated and stable cardiovascular disease may participate
* Have plasma total cholesterol > 200 mg/dL or plasma triglycerides > 200 mg/dL
* Have a calculated glomerular filtration rate (GFR) =< 30 mL/min/1.73 m^2
* Are not free of unstable angina, arrhythmia, or severe systemic disease that would make moderate intensity exercise participation unsafe
* Have any contra-indications to magnetic resonance (MR) examination such as allergy to MRI contrast media (gadolinium-DTPA [gadopentetate dimeglumine]), metallic foreign objects within the body, orbital metal, cerebral aneurysm clip, pacemaker, defibrillator, neurostimulator, any other medical metallic implant, claustrophobia, inability to lie flat for 30 minutes, and weight exceeding 300 pounds; if an MR contraindication is discovered during scanning that was overlooked during the screening process, the procedure will be stopped immediately and the subject will be removed from the scanner
* Are receiving any form of renal replacement therapy or have a calculated glomerular filtration rate (GFR) < 30 mL/min/1.75 m²; results of serum creatinine testing will be reviewed for calculation of glomerular filtration rate (GFR); patients without a serum creatinine level drawn within the prior 3 months will have this drawn upon enrollment
* Have uncontrolled hypertension and resting blood pressure exceeding 140/80 mmHg
* In addition, subjects with any contraindications to exercise testing according to American Heart Association guidelines will not be enrolled; nonetheless, the cardiovascular magnetic resonance (CMR) cardiologist supervising the research portion of the exam will also evaluate each subject for evidence of any contra-indications; the absolute contra-indications include acute myocardial infarction, high-risk unstable angina, uncontrolled cardiac arrhythmias, active endocarditis, symptomatic severe aortic stenosis, decompensated symptomatic heart failure, acute pulmonary embolus or pulmonary infarction, acute non-cardiac disorder that may be aggravated by exercise, acute myocarditis or pericarditis, physical disability that would preclude safe and adequate test performance, and inability to provide consent; the relative contra-indications include left main coronary stenosis, moderate stenotic valvular heart disease, electrolyte abnormalities, tachyarrhythmias or bradyarrhythmias, atrial fibrillation with uncontrolled ventricular rate, hypertrophic cardiomyopathy, and high-degree atrioventricular node block; subjects with uncontrolled hypertension and resting blood pressure exceeding 140/80 mmHg will be excluded

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate (bpm) | Up to 7 months post ADT initiation
Maximal rate of oxygen consumption | Up to 7 months post ADT initiation
Cardiac muscle mass | Up to 7 months post ADT initiation
Ventricular performance assessed by cardiac stress MRI | Up to 7 months post ADT initiation
Myocardial perfusion reserve assessed by cardiac stress MRI | Up to 7 months post ADT initiation
Skeletal muscle energetics assessed by PMRS | Up to 7 months post ADT initiation

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu